CLINICAL TRIAL: NCT02040415
Title: A Multicenter, Randomized, Double-blinded, Parallel, Active-controlled, Phase Lll Clinical Trial to Evaluate the Efficacy and Safety of DW-1030 and Eperisone HCl in Acute Back Pain Patients
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of DW-1030 and Eperisone HCl in Acute Back Pain Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW-1030_301
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Acute Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- DW-1030(eperisone HCl) (Experimental): DW-1030(eperisone HCl) 75mg BID
  Interventions: Drug: DW-1030(eperisone HCl) 75mg; Drug: Placebo drug of Myonal Tab.
- Myonal Tab.(eperisone HCl) (Active Comparator): Myonal Tab.(eperisone HCl) 50mg TID
  Interventions: Drug: Myonal Tab.(eperisone HCl) 50mg; Drug: Placebo drug of DW-1030

INTERVENTIONS:
Drug: DW-1030(eperisone HCl) 75mg
  Arms: DW-1030(eperisone HCl)
Drug: Myonal Tab.(eperisone HCl) 50mg
  Arms: Myonal Tab.(eperisone HCl)
Drug: Placebo drug of DW-1030
  Arms: Myonal Tab.(eperisone HCl)
Drug: Placebo drug of Myonal Tab.
  Arms: DW-1030(eperisone HCl)

SUMMARY:
The purpose of this clinical study is to determine whether or not DW-1030 is not inferior to eperisone HCl in efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult males/Females aged over 18 years
* Patients with symptom of Acute skeletomuscle myospasm and Back pain
* Patients with Pain VAS Value over 40 mm in Visit 2
* Subjects who voluntarily or legal guardian agreed with written consent

Exclusion Criteria:

* Patients with Back pain caused by spinal spondylosis, spinal stenosis, fractures, cancer, severe arthritis, osteoporosis, sciatica, infection
* Muscular patients such as myositis, muscular atrophy disease, increased muscle tone, myasthenia gravis
* Patients who had taken invasive procedures such as epidural injections or spinal stimulation to cure the back pain within 6 months from the screening point
* Patients who had taken passive physical therapy or ionphoresis within 12 hours from the screening point
* Patients with severe GI tract disorder, heart disease, hypertension
* Patients who had taken NSAIDS within 24hours from the screening point

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Changes of Finger-to-Floor Distance(FFD) compared to baseline 7days after administration | 1, 3, 7 day

SECONDARY OUTCOMES:
Changes of 100mm Pain VAS | -3, 1, 3, 7 day
Oswestry Disability Index (ODI) | 1, 3, 7 day
Physician's Global Assessment | 7 day
The number of using rescue drugs and the total amount | 1, 3, 7 days